CLINICAL TRIAL: NCT00940654
Title: The Fever and Antipyretic in Critically Illness Evaluation Study
Acronym: FACE
Status: Completed | Type: Observational
Sponsor: Japanese Society of Intensive Care Medicine (Other)
Responsible Party: Japanese Society of Intensive Care Medicine, Japanese Society of Intensive Care Medicine
Other Study IDs: JSICM&KSCCM FACE
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2009-09

CONDITIONS: Fever; Hyperthermia
Keywords: Fever; Antipyretic; Infection; Mortality; Cooling; Non steroid anti inflammatory drugs; Acetaminophen; Steroid; ICU; Intensive care; Critically ill
MeSH Terms: conditions — Fever; Hyperthermia; Infections; Critical Illness | interventions — Acetaminophen; Steroids; Bro protein, Drosophila

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with fever
  Interventions: Other: Antipyretic therapy
- Patients without any fever

INTERVENTIONS:
Other: Antipyretic therapy — External cooling;Internal cooling;Non steroid anti inflammatory drugs; Acetaminophen; Steroid
  Other Names: External cooling; Internal cooling; Non steroid anti inflammatory drugs; Acetaminophen; Steroid; Others
  Groups: Patients with fever

SUMMARY:
The purpose of this multination multicenter observational study is to determine the impact of fever and antipyretic on outcomes in critically ill patients.

DETAILED DESCRIPTION:
Fever is common in critically ill patients.Antipyretic therapy for fever is routinely performed in intensive care.There are studies to assess the relationship between fever and mortality in non-neurological ICU. However, all of them did not have any information of antipyretic therapy. There are two small, single center RCT, which suggested a potential risk for antipyretic therapy. Thus, a large RCT might be ethically difficult.

It is unfortunate that there is not enough information on how the investigators should control body temperature in non-neurological critically ill patients, because fever is a very common physiological abnormality in this cohort. From the beginning, it would, therefore, be desirable to understand several aspects of fever and antipyretic therapy in ICU patients, as 1)How often fever occurs in our ICUs, 2)To what degree fever is independently associated with mortality?, 3)How often antipyretic therapy is prescribed?, 4)How effectively antipyretic can decrease temperature?, 5)How different is lowering temperature with medications compared with cooling?, 6)To what degree antipyretic is independently associated with mortality?

Thus, the investigators plan to address these questions by conducting a multi-national multi-center prospective observational trial, named "The Fever and Antipyretic in Critically illness evaluation study" (The FACE study)

ELIGIBILITY:
Inclusion Criteria:

* Adult non-neurological critically ill patients (20 years old or older).
* ICU patients expected to require intensive care for more than 48 hour.

Exclusion Criteria:

* Patients with brain injury (suspected or proven)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult non-neurological critically ill patients required intensive care for more than 48 hour.
Sampling Method: Probability Sample
Enrollment: 1426 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
28 days mortality | 28days after ICU admission

SECONDARY OUTCOMES:
ICU free days at 28 days | 28 days after ICU admission
Hospital free days at 28 days | 28 days
Ventilator free days at 28 days | 28 days at ICU admission
Renal replacement therapy free days at 28 days | 28 days at ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Younsuck Koh, M.D. PhD, Study Chair — Korean Society of Critical Care Medicine; Masaji Nishimura, M.D. PhD, Study Chair — Japanese Society of Intensive Care Medicine; Jae Yeol Kim, M.D., Principal Investigator — Korean Society of Critical Care Medicine; Gee Young Suh, M.D., Principal Investigator — Korean Society of Critical Care Medicine; Moritoki Egi, M.D., Principal Investigator — Japanese Society of Intensive Care Medicine
Locations (2):
- The Japanese Society of Intensive Care Medicine, Bunkyo-ku, Tokyo, Japan
- Korean Society of Critical Care Medicine, Songpa-gu, Seoul, South Korea

REFERENCES:
- [Derived] Lee BH, Inui D, Suh GY, Kim JY, Kwon JY, Park J, Tada K, Tanaka K, Ietsugu K, Uehara K, Dote K, Tajimi K, Morita K, Matsuo K, Hoshino K, Hosokawa K, Lee KH, Lee KM, Takatori M, Nishimura M, Sanui M, Ito M, Egi M, Honda N, Okayama N, Shime N, Tsuruta R, Nogami S, Yoon SH, Fujitani S, Koh SO, Takeda S, Saito S, Hong SJ, Yamamoto T, Yokoyama T, Yamaguchi T, Nishiyama T, Igarashi T, Kakihana Y, Koh Y; Fever and Antipyretic in Critically ill patients Evaluation (FACE) Study Group. Association of body temperature and antipyretic treatments with mortality of critically ill patients with and without sepsis: multi-centered prospective observational study. Crit Care. 2012 Feb 28;16(1):R33. doi: 10.1186/cc11211. PMID 22373120
- See also: JSICM — http://www.jsicm.org/en/